CLINICAL TRIAL: NCT00174564
Title: A Multicentre Phase II Trial of Gemcitabine and Oxaliplatin (GEMOX) in Patients With Biliary Tract Cancer
Brief Title: EXIBIT: Oxaliplatin in Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C_8552
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Biliary Tract Neoplasms
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Oxaliplatin

INTERVENTIONS:
Drug: oxaliplatin

SUMMARY:
The primary objective is to evaluate the efficacy of the GEMOX treatment as 1st line therapy in patients with advanced biliary tract cancer based on response rate measured by the RECIST unidimensional criteria.

Secondary objectives are : Progression free survival, overall survival and safety.

ELIGIBILITY:
* Histologically proven, locally advanced or metastatic carcinoma of the biliary tract (gallbladder, intrahepatic bile ducts, extrahepatic bile ducts, ampula of Vater)
* For intrahepatic bile ducts, if the diagnosis of biliary tract origin is not evident by imaging or surgical exploration, and so equivalent to liver metastasis with unknown primary site, inclusion is possible if:

  * unknown primary after an exhaustive search for the primary site (chest radiography- , thoracic and abdomino pelvic CT scan, colonoscopy, oesogastroduodenal endoscopy, PSA determination for men or mammography for women, and PET scan if possible).
  * histological examination compatible with adenocarcinoma of bile ducts with the immunostaining expression of cytokeratin : 7+, 20- and 19 +. (Shimonishi, 2000 ^22)
* No prior chemotherapy for advanced disease (first line)
* No radiation therapy within 4 weeks prior to the first gemcitabine administration.
* Unidimensionally measurable disease.
* For female patient of childbearing potential, neither pregnant nor breastfeeding, and under active contraception
* No known allergy to one of the study drugs
* No prior malignancy
* No CNS metastases
* No peripheral neuropathy > grade 2
* ECOG PS <=2
* ANC > 1.5 X 10^9 /L
* Platelets > 100 X 10^9 /L
* Creatinine < 1.5 x ULN
* SGPT (ALT) < 5 x ULN
* Bilirubin < 2.5 x ULN (patients with jaundice or evidence of bile duct obstruction and in whom the biliary tree can be decompressed by endoscopic percutaneous endoprothesis, with subsequent reduction in bilirubin < 2.5 x ULN will be eligible for the study).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2003-04; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
To evaluate response rate according to RECIST criteria

SECONDARY OUTCOMES:
To evaluate the progression-free survival in the ITT population
To investigate safety using NCI-CTC criteria version 2

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Aussel, Study Director — Sanofi